CLINICAL TRIAL: NCT06979869
Title: Investigating Multigene Methylation Dynamics in Treatment Response Surveillance for Esophageal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20252117-F-1
Record Dates: First submitted 2025-04-23; First posted 2025-05-20 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group one: Esophageal cancer patients undergoing primary surgical treatment
  Interventions: Other: Multi-gene methylation testing
- Group two: Esophageal cancer patients undergoing surgery following neoadjuvant therapy
  Interventions: Other: Multi-gene methylation testing
- Group three: Esophageal cancer patients undergoing active surveillance following neoadjuvant therapy
  Interventions: Other: Multi-gene methylation testing
- Group four: Esophageal cancer patients undergoing definitive chemoradiotherapy with or without immunotherapy
  Interventions: Other: Multi-gene methylation testing

INTERVENTIONS:
Other: Multi-gene methylation testing — Undergo multi-gene methylation testing in blood during follow-up
  Groups: Group one
Other: Multi-gene methylation testing — Undergo multi-gene methylation testing in blood during follow-up
  Groups: Group two
Other: Multi-gene methylation testing — Undergo multi-gene methylation testing in blood during follow-up
  Groups: Group three
Other: Multi-gene methylation testing — Undergo multi-gene methylation testing in blood during follow-up
  Groups: Group four

SUMMARY:
The primary objective is to determine whether pretreatment-to-posttreatment changes in circulating multigene methylation levels correlate with objective response rates (ORR) assessed by contrast-enhanced CT/MRI and levels of serum tumor markers. Secondary endpoints include: (a) time-dependent association between methylation fluctuation patterns and progression-free survival (PFS), (b) comparative diagnostic accuracy of methylation indices versus conventional biomarkers, and (c) feasibility of using methylation thresholds to guide adaptive therapy modification.

ELIGIBILITY:
Inclusion Criteria:

Age at initial diagnosis: 18-75 years (inclusive) Confirmed diagnosis: Histologically proven esophageal carcinoma with complete medical records, including (a) definitive pathological diagnosis report, (b) TNM staging per AJCC 8th edition criteria Cancer history: No prior malignancies at other anatomical sites (excluding cured non-melanoma skin cancers/carcinoma in situ) Metastasis status: Radiologically confirmed absence of distant metastases in liver, lungs, or other organs via contrast-enhanced CT/MRI and whole-body bone scan within 4 weeks before enrollment Treatment-naïve status: No previous exposure to (i) esophageal resection surgery, (ii) systemic chemotherapy, (iii) thoracic radiation therapy (>10 Gy), or (iv) PD-1/PD-L1 immune checkpoint inhibitors

Exclusion Criteria:

Life expectancy <6 months (as assessed by ECOG score ≥4 or Palliative Performance Scale ≤30%) Cognitive/psychiatric conditions: a. Legally incapacitated individuals without legal guardians, b. Active psychotic disorders (e.g., schizophrenia, bipolar disorder) or dementia (MMSE score <24) Investigator-determined exclusions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Multi-gene methylation levels | Group one: Preoperative, 1 week, 1 month, 3 months, 6 months, 1 year, 1.5 years, 2 years, 3 years, 4 years, and 5 years postoperatively.
Multi-gene methylation levels | Group two: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and postoperatively at 1 week, 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
Multi-gene methylation levels | Group three: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and post-neoadjuvant therapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
Multi-gene methylation levels | Group four: pre-definitive chemoradiotherapy baseline, and post-definitive chemoradiotherapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.

SECONDARY OUTCOMES:
Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) | Group one: Preoperative, 1 week, 1 month, 3 months, 6 months, 1 year, 1.5 years, 2 years, 3 years, 4 years, and 5 years postoperatively.
  Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) results will be extracted from historical medical records, with test dates typically ranging from baseline (within 3 months pre-enrollment) to follow-up intervals aligned with standard clinical practice (e.g., every 3-6 months post-treatment). These time points may not synchronize with the methylation assessment schedule.
Imaging Examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) | Group one: Preoperative, 1 week, 1 month, 3 months, 6 months, 1 year, 1.5 years, 2 years, 3 years, 4 years, and 5 years postoperatively.
  Imaging examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Endoscope | Group one: Preoperative, 1 week, 1 month, 3 months, 6 months, 1 year, 1.5 years, 2 years, 3 years, 4 years, and 5 years postoperatively.
  Endoscoping results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) | Group two: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and postoperatively at 1 week, 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) results will be extracted from historical medical records, with test dates typically ranging from baseline (within 3 months pre-enrollment) to follow-up intervals aligned with standard clinical practice (e.g., every 3-6 months post-treatment). These time points may not synchronize with the methylation assessment schedule.
Imaging Examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) | Group two: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and postoperatively at 1 week, 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Imaging examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Endoscope | Group two: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and postoperatively at 1 week, 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Endoscoping results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) | Group three: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and post-neoadjuvant therapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) results will be extracted from historical medical records, with test dates typically ranging from baseline (within 3 months pre-enrollment) to follow-up intervals aligned with standard clinical practice (e.g., every 3-6 months post-treatment). These time points may not synchronize with the methylation assessment schedule.
Imaging Examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) | Group three: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and post-neoadjuvant therapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Imaging examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Endoscope | Group three: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and post-neoadjuvant therapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Endoscoping results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) | Group four: pre-definitive chemoradiotherapy baseline, and post-definitive chemoradiotherapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) results will be extracted from historical medical records, with test dates typically ranging from baseline (within 3 months pre-enrollment) to follow-up intervals aligned with standard clinical practice (e.g., every 3-6 months post-treatment). These time points may not synchronize with the methylation assessment schedule.
Imaging Examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) | Group four: pre-definitive chemoradiotherapy baseline, and post-definitive chemoradiotherapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Imaging examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Endoscope | Group four: pre-definitive chemoradiotherapy baseline, and post-definitive chemoradiotherapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Endoscoping results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Gansu Wuwei Cancer Hospital, Wuwei, Gansu
  - Cancer Hospital Affiliated to Shantou University Medical College, Shantou, Guangdong
  - Zhaoqing Gaoyao District People's Hospital, Zhaoqing, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tangdu Hospital, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Yan'an University, Yan’an, Shaanxi
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - General Hospital of Western Theater Command, People's Liberation Army (PLA), Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided